CLINICAL TRIAL: NCT03248505
Title: Immediate Effects of Conventional TENS and Burst TENS Combined With Cryotherapy in the Non-specific Low Back Pain
Brief Title: Cryotherapy and TENS on Low Back Pain
Acronym: CTLBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Professor of Physiotherapy, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TENS_LBP
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation; Cryotherapy; Ice

STUDY DESIGN:
Intervention Model Description: 3x6
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo TENS (Placebo Comparator): TENS unit turned on, but with zero amplitude.
  Interventions: Other: Placebo TENS
- Conventional TENS (Experimental): Symmetrical biphasic pulsed current, with frequency of 100 Hz, pulse duration of 100 micro-seconds and sensory-level amplitude.
  Interventions: Device: Conventional TENS
- Burst TENS (Experimental): Carrier frequency of 100 Hz burst-modulated at 4Hz, pulse duration of 200 micro-seconds and motor-level amplitude.
  Interventions: Device: Burst TENS
- Cryotherapy (Experimental): 1,5 Kg crushed ice pack
  Interventions: Other: Cryotherapy
- Burst TENS + Cryotherapy (Experimental): Carrier frequency of 100 Hz burst-modulated at 4Hz, pulse duration of 200 micro-seconds and motor-level amplitude plus an ice pack of 1,5 Kg.
  Interventions: Device: Burst TENS + Cryotherapy
- Conventional TENS + Cryotherapy (Experimental): Symmetrical biphasic pulsed current, with frequency of 100 Hz, pulse duration of 100 micro-seconds and sensory-level amplitude plus an ice pack of 1,5 Kg.
  Interventions: Device: Conventional TENS + Cryotherapy

INTERVENTIONS:
Device: Conventional TENS — Transcutaneous Electrical Nerve Stimulation (frequency of 100 Hz, pulse duration of 100 micro-seconds and sensory-level amplitude) with two electrodes in each side of the lumbar spinal.
  Other Names: Transcutaneous Electrical Nerve Stimulation
  Arms: Conventional TENS
Device: Burst TENS — Burst-modulated TENS with carrier frequency of 100 Hz, burst-modulated at 4Hz, pulse duration of 200 micro-seconds and motor-level amplitude.
  Other Names: Burst-modulated TENS
  Arms: Burst TENS
Other: Cryotherapy — 1,5 Kg of crushed ice pack on lumbar spine.
  Other Names: Ice
  Arms: Cryotherapy
Device: Burst TENS + Cryotherapy — Burst-modulated TENS with carrier frequency of 100 Hz, burst-modulated at 4Hz, pulse duration of 200 micro-seconds and motor-level amplitude plus 1,5 Kg of crushed ice pack on lumbar spine.
  Other Names: Burst-modulated TENS and Ice
  Arms: Burst TENS + Cryotherapy
Device: Conventional TENS + Cryotherapy — Transcutaneous Electrical Nerve Stimulation (frequency of 100 Hz, pulse duration of 100 micro-seconds and sensory-level amplitude) plus s 1,5 Kg of crushed ice pack on lumbar spine.
  Other Names: Transcutaneous Electrical Nerve Stimulation + Ice
  Arms: Conventional TENS + Cryotherapy
Other: Placebo TENS — TENS device turned on, but with zero amplitude.
  Other Names: Placebo
  Arms: Placebo TENS

SUMMARY:
This study aim analyze the immediate effects of conventional transcutaneous electrical nerve stimulation (TENS) and Burst TENS combined or not with cryotherapy in patients with non-specific low back pain.

All subjects will be submitted to an evaluation of the painful sensation, through the numerical rating scale, and pain threshold, through algometry, before, immediately after the intervention and 25 minutes after.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 50 years;
* Have chronic non-specific low back pain.

Exclusion Criteria:

* Serious spinal pathologies (fractures, tumors, and inflammatory pathologies such as ankylosing spondylitis);
* Nerve root compromise (disc herniation and spondylolisthesis with neurological compromise, spinal stenosis, and others);
* Fibromyalgia
* Corticosteroid treatment in the previous two weeks;
* Antiinflammatory treatment in the previous 24 hours;
* Contraindications to the use of Kinesio Taping (allergy or intolerance);
* Score of three or less on Visual Analogue Scale of the first day;
* Pregnancy;
* Ice allergy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-05-29 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Painful sensation | Evaluation of pain sensation 25 minutes after the application of the intervention.
  Pain sensation measured by pain numerical rating scale

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: Undecided